CLINICAL TRIAL: NCT06222229
Title: Multicentre, Randomized, Clinical Trial in Children With Mild Ankle Sprain: Bandaging vs. no Immobilization
Brief Title: Mild Ankle Sprain Treatment: Functional Bandaging vs. no Immobilization
Acronym: PED_HUIL0124
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Universitario Infanta Leonor (Other)
Responsible Party: Principal Investigator, ÁNGEL PUEYO, MD, MSc, Pediatric Specialist Physician, Hospital Universitario Infanta Leonor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PED_HUIL0124
Record Dates: First submitted 2024-01-03; First posted 2024-01-24 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Primary Disease or Condition Being Studied in the Trial or the Focus of the Study Mild Ankle Sprain
Keywords: Ankle; Sprain
MeSH Terms: conditions — Sprains and Strains

STUDY DESIGN:
Intervention Model Description: Randomization sequence was created using the Epidat 4.2 software, ensuring allocation concealment, with a single, constant 1:1 allocation ratio
Masking Description: Due to the nature of the intervention, it will not be feasible to mask the received treatment at the time of care. Additionally, masking of the treatment group during clinical reviews will not be attainable, as some collected variables will be inherently related to the intervention itself. The data analyst specialist will also be unblinded to the group assignments.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No-bandaging group (Experimental): Only general measures will be recommended without the use of external support devices.
  Interventions: Other: Control
- Bandaging group (Active Comparator): functional bandage for 5 days and general measure.
  Interventions: Other: Control; Procedure: Functional bandage

INTERVENTIONS:
Other: Control — All patients included in the study, both in the non-bandaging group and in the bandaging group, will receive a series of general measures as a recommendation, consisting of the following:
  * Administration of anti-inflammatory drugs as ibuprofen at 7.5 mg/kg/8 hours for 2-3 days. If pain continues, recommendation of paracetamol 15 mg/kg 4 hours after ibuprofen.
  * Application of local ice for a maximum of 10 minutes as required.
  * Elevation of the affected limb when resting.
  * Early mobilization and load according to tolerance, using crutches if required.
  * Sports rest at least for one week or until the patient is able to walk without pain, with gradual incorporation according to tolerance. During the following year, use of elastic ankle brace for sports activities.
  The control group will not receive any special intervention.
Procedure: Functional bandage — The functional bandage will consist of a standardized wrapping in several phases. First, with 6 mm silk tape, open anchors were placed in the distal region of the metatarsals of the foot and in the middle third of the affected leg. Next, a strip of tape was applied in stirrup fashion, starting from the proximal anchor and exerting pressure cranially on the side of the affected ligament. This support was interspersed three times with another strip of tape, starting from the foot anchor and wrapping behind the ankle. Once complete, it was covered with a 7.5 cm Tensoplast spiral bandage, taking care to apply gentle pressure. The emergency nurses underwent dual training, consisting of an instructional video and a half-hour practical session. Reminder posters were also displayed in the technique box where such procedures are typically performed.
  As the control group, general measures will be recommended
  Arms: Bandaging group

SUMMARY:
Ankle sprains represent a prevalent pathology among the pediatric population that can result in residual effects when treated incorrectly. However, there is a lack of scientific studies defining the most appropriate therapeutic approach. The hypothesis is that patients treated solely with general measures, without external device support, experience a faster recovery compared to those treated with ankle immobilization. A clinical trial will be carried out by randomly assigning patients to either the functional bandaging group or the control group (general measures only). Prospective follow-up will be carried out by a online survey send by SMS, checking the functionality of the injured ankle using 'the Oxford Ankle Foot Questionnaire for Children (OxAFQ-C)', in addition to pain control and patient satisfaction with the treatment.

DETAILED DESCRIPTION:
Study Design: A randomized, parallel, open-label, multi-center clinical trial will be conducted at 3 intermediate-complexity hospitals. The study received approval from the center's ethics committee.

Procedure: Every patient presenting with ankle trauma will undergo assessment by the attending physician in the emergency department. The collaborating researchers of the different hospitals will participate in patient enrollment. In cases of grade I or mild sprains, patients and their guardians will be invited to participate in the study after a thorough explanation of the study's purpose and procedures. The severity of the sprain will be assessed using The West Point Ankle Grading System. Adequate analgesia will be ensured during the emergency department consultation.

Upon agreeing to participate in the study and signing the informed consent, randomization and assignment to either the control group or intervention group (receiving a bandage applied by nursing) will take place before the final discharge from the emergency department. The discharge report will specify the standardized treatment based on the assigned group. The attending physician will complete a physical study-specific record and will store the signed informed consent in a designated folder within the pediatric emergency department. The researcher in charge of each center will enter demographic data and variables obtained in the emergency department into a database hosted in the REDcap software. The data of the recruited patients should be entered in the REDcap database at least twice per week. The principal investigator or collaborators will review this REDcap database daily to check the recruited patients and prepare the SMS with the online survey to be sent. A coded patient number and the date of emergency care will be included in a database hosted in the center's electronic repository to determine the timing of follow-up. The SMS will be sent using the SMS sending system of the coordinating hospital of the study.

At 7, 14, and 30 days, the guardians of the patients will receive a SMS with a link that will direct them to the REDcap online survey. In case of no response to the initial attempt, another attempt will be made the following day, and, if no response is received in 48 hours, a telephone call will be made to the patients' guardians. Non-response at 72 hours will be recorded as a loss.

The data from the REDcap electronic database will be periodically reviewed by the principal investigator to monitore data entry and look for possible adverse effect.

Statistical Analysis: The sample size will be calculated assuming a difference of more than 10 points in the OXAFQ-C percentage scale value, estimating a standard deviation of 15, due to a previous study. Comparing two independent means with a bilateral test and a balanced random allocation (Group 1 size/Group 2 size ratio = 1), with a type I error of 5% (alpha risk) and a power of 80% (1-beta risk), and assuming a dropout of 30%, the calculated sample size will be 112 patients (56 in each group) for superiority analysis or 90 patients (45 in each group) for non-inferiority analysis.

Categorical variables will be described using percentages, and continuous variables will be presented as mean and standard deviation (SD) if normally distributed (Kolmogorov-Smirnov and/or Shapiro-Wilks) or as medians and interquartile ranges otherwise. Bivariable analysis of categorical variables will be performed using the Chi-square test or Fisher's exact test, and that of continuous variables will be done using the Student's T-test or its non-parametric equivalents.

Both intention-to-treat and per-protocol analyses will be conducted, assuming that some patients in the control group will use ankle support against recommendations. Finally, a non-inferiority analysis will be performed between both groups for both the primary variable and the degree of pain according to the visual analog scale (VAS) at different follow-ups.

All statistical tests will be considered with a significance level of 5%. The analysis will be conducted using the R software.

Missing Data:For all patients who do not complete at least two follow-ups, the electronic medical records of all public centers in the province where the study is conducted will be reviewed through the electronic Horus program to verify the absence of relevant adverse effects or diagnostic changes. Anyway, a worst-case scenario strategy will be used in the statistical analysis to assess the losses.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of grade I ankle sprain.
* Patients aged between 5 and 16 years.
* Less than 72 hours of evolution.
* Informed consent signed by guardians

Exclusion Criteria:

* Penetrating trauma.
* Associated fracture.
* Consultation more than 72 hours after the trauma.
* Developmental disorders (cerebral palsy, previous gait disorders, autism, etc.).
* Previous or concurrent disease that involves an increased risk of fractures (osteoporosis, bone diseases, etc).
* Previous ankle pathology.
* Impossibility of telephone contact

Ages: 5 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Percentage score on the Oxford Ankle and Foot Questionare for Children (OXAFQ-C) | at 5, 14 and 30 days.
  It is a questionnaire validated in pediatric population to determine the functionality of the ankle and/or foot in patients with pathology at this level. It consists of a survey in which 14 items belonging to three different spheres are collected: physical, social/daily activities and emotional. Each item is scored on a frequency scale: never (4), rarely (3), sometimes (2), frequently (1), always (0). The higher the score, the better the functionality. This scale can also be transformed into a percentage scale, being 100% the maximum score.
Intensity of pain | at the emergency department and at 5, 14 and 30 days.
  intensity of pain felt by the patient, assessed subjectively on an ordinal scale, with 0 being no pain at all and 10 the maximum pain possible.
recurrence of ankle sprain | at 5, 14 and 30 days.
  dichotomous variable reflecting the presence of new ankle sprains.

SECONDARY OUTCOMES:
patient satisfaction with emergency department care | after 5 days
  assessed subjectively on an ordinal scale, being 0 being the worst punctuation and 10 being the best.
Patient satisfaction with the treatment received. | after 5 days
  assessed subjectively on an ordinal scale, being 0 being the worst punctuation and 10 being the best.
Patient satisfaction with functional evolution. | after 30 days
  assessed subjectively on an ordinal scale, being 0 being the worst punctuation and 10 being the best.
Presence of functional bandaging complications | after 5 days
  dichotomous variable (yes/no).
Tolerance of the functional bandage | after 5 days
  ordinal scale (very bad, bad, average, good and very good).
Use of crutches | after 5 days
  dichotomous variable (yes/ no)
Days on crutches | after 5 days
  quantitative variable (days)
Days of use of anti-inflammatory drugs | after 5 days
  quantitative variable (days)
Days with pain | at 5, 14 and 30 days.
  quantitative variable (days)
Use of ankle brace | at 5, 14 and 30 days.
  dichotomous variable (yes/ no)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Infanta Leonor, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Saki F, Yalfani A, Fousekis K, Sodejani SH, Ramezani F. Anatomical risk factors of lateral ankle sprain in adolescent athletes: A prospective cohort study. Phys Ther Sport. 2021 Mar;48:26-34. doi: 10.1016/j.ptsp.2020.12.009. Epub 2020 Dec 16. PMID 33352395
- [Result] Waterman BR, Owens BD, Davey S, Zacchilli MA, Belmont PJ Jr. The epidemiology of ankle sprains in the United States. J Bone Joint Surg Am. 2010 Oct 6;92(13):2279-84. doi: 10.2106/JBJS.I.01537. PMID 20926721
- [Result] Wiersma AJ, Brou L, Fields SK, Comstock RD, Kerr ZY. Epidemiologic comparison of ankle injuries presenting to US emergency departments versus high school and collegiate athletic training settings. Inj Epidemiol. 2018 Sep 3;5(1):33. doi: 10.1186/s40621-018-0163-x. PMID 30175385
- [Result] Czajka CM, Tran E, Cai AN, DiPreta JA. Ankle sprains and instability. Med Clin North Am. 2014 Mar;98(2):313-29. doi: 10.1016/j.mcna.2013.11.003. Epub 2014 Jan 10. PMID 24559877
- [Result] Altomare D, Fusco G, Bertolino E, Ranieri R, Sconza C, Lipina M, Kon E, Marcacci M, Bianchini L, Di Matteo B. Evidence-based treatment choices for acute lateral ankle sprain: a comprehensive systematic review. Eur Rev Med Pharmacol Sci. 2022 Mar;26(6):1876-1884. doi: 10.26355/eurrev_202203_28333. PMID 35363336
- [Result] Delahunt E, Bleakley CM, Bossard DS, Caulfield BM, Docherty CL, Doherty C, Fourchet F, Fong DT, Hertel J, Hiller CE, Kaminski TW, McKeon PO, Refshauge KM, Remus A, Verhagen E, Vicenzino BT, Wikstrom EA, Gribble PA. Clinical assessment of acute lateral ankle sprain injuries (ROAST): 2019 consensus statement and recommendations of the International Ankle Consortium. Br J Sports Med. 2018 Oct;52(20):1304-1310. doi: 10.1136/bjsports-2017-098885. Epub 2018 Jun 9. PMID 29886432
- [Result] Gaddi D, Mosca A, Piatti M, Munegato D, Catalano M, Di Lorenzo G, Turati M, Zanchi N, Piscitelli D, Chui K, Zatti G, Bigoni M. Acute Ankle Sprain Management: An Umbrella Review of Systematic Reviews. Front Med (Lausanne). 2022 Jul 7;9:868474. doi: 10.3389/fmed.2022.868474. eCollection 2022. PMID 35872766
- [Result] Lacerda D, Pacheco D, Rocha AT, Diniz P, Pedro I, Pinto FG. Current Concept Review: State of Acute Lateral Ankle Injury Classification Systems. J Foot Ankle Surg. 2023 Jan-Feb;62(1):197-203. doi: 10.1053/j.jfas.2022.08.005. Epub 2022 Aug 18. PMID 36184447
- [Result] Maughan K.L., Jackson J. Ankle sprain in adults: Evaluation and diagnosis. En: UpToDate. 2023.
- [Result] Maughan K.L., Jackson J. Ankle sprain in adults: Management. En 2023.
- [Result] Green T, Willson G, Martin D, Fallon K. What is the quality of clinical practice guidelines for the treatment of acute lateral ankle ligament sprains in adults? A systematic review. BMC Musculoskelet Disord. 2019 Aug 31;20(1):394. doi: 10.1186/s12891-019-2750-6. PMID 31470826
- [Result] Jones P, Lamdin R, Dalziel SR. Oral non-steroidal anti-inflammatory drugs versus other oral analgesic agents for acute soft tissue injury. Cochrane Database Syst Rev. 2020 Aug 12;8(8):CD007789. doi: 10.1002/14651858.CD007789.pub3. PMID 32797734
- [Result] Derry S, Moore RA, Gaskell H, McIntyre M, Wiffen PJ. Topical NSAIDs for acute musculoskeletal pain in adults. Cochrane Database Syst Rev. 2015 Jun 11;2015(6):CD007402. doi: 10.1002/14651858.CD007402.pub3. PMID 26068955
- [Result] Tran K, Argaez C. External Supports for the Treatment of Ankle Sprain: A Review of Clinical Effectiveness [Internet]. Ottawa (ON): Canadian Agency for Drugs and Technologies in Health; 2020 May 1. Available from http://www.ncbi.nlm.nih.gov/books/NBK563450/ PMID 33112532
- [Result] Gogate N, Satpute K, Hall T. The effectiveness of mobilization with movement on pain, balance and function following acute and sub acute inversion ankle sprain - A randomized, placebo controlled trial. Phys Ther Sport. 2021 Mar;48:91-100. doi: 10.1016/j.ptsp.2020.12.016. Epub 2020 Dec 23. PMID 33401232
- [Result] Bleakley CM, O'Connor SR, Tully MA, Rocke LG, Macauley DC, Bradbury I, Keegan S, McDonough SM. Effect of accelerated rehabilitation on function after ankle sprain: randomised controlled trial. BMJ. 2010 May 10;340:c1964. doi: 10.1136/bmj.c1964. PMID 20457737
- [Result] Iammarino K, Marrie J, Selhorst M, Lowes LP. EFFICACY OF THE STRETCH BAND ANKLE TRACTION TECHNIQUE IN THE TREATMENT OF PEDIATRIC PATIENTS WITH ACUTE ANKLE SPRAINS: A RANDOMIZED CONTROL TRIAL. Int J Sports Phys Ther. 2018 Feb;13(1):1-11. PMID 29484236